CLINICAL TRIAL: NCT00125203
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Safety and Efficacy of Botulinum Toxin Type B (Myobloc) in Sialorrhea in Amyotrophic Lateral Sclerosis
Brief Title: Study of Myobloc in the Treatment of Sialorrhea (Drooling) in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: ALS Association (Other); University of Kansas (Other); Carolinas MDA Neuromuscular/ALS Center-Carolinas Medical System (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB-IND 11090
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Sialorrhea
Keywords: ALS; Lou Gehrig's Disease; Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Sialorrhea; Hypersalivation; Excessive Drooling; Myobloc; botulinum toxin type B; Clostridium botulinum B toxin; botulinum B toxin; botulinum neurotoxin B; NeuroBloc
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Sialorrhea; Motor Neuron Disease | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Botulinum toxin type B (Myobloc)
Procedure: Injection of salivary glands

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Myobloc in ALS patients who are having excessive drooling.

The primary goal of the study is to determine if the patient perceives a benefit from the Myobloc in controlling excessive drooling.

DETAILED DESCRIPTION:
The secondary goals of this study are to:

* determine the safety of bilateral injections of Myobloc into the parotid and submandibular glands as an effort to control sialorrhea;
* determine by objective measures if the Myobloc injection decreases the saliva produced;
* determine caregiver perceived benefit from Myobloc injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite ALS based on current World Federation of Neurology criteria
* Between the ages of 21-85, inclusive
* Sialorrhea refractory to treatment with at least two anticholinergic medications OR has been intolerant of anticholinergic medications due to side effects
* Capable of giving informed consent
* Must be able to attend all study visits

Exclusion Criteria:

* Patient has any uncontrolled significant medical, psychiatric or neurological disease (other than ALS) over the past 30 days
* History of ongoing substance abuse
* History of non-compliance with treatment in other experimental protocols
* Cannot provide informed consent or comply with evaluation procedures
* Has received any form of botulinum toxin in the past for any indication
* Women who are pregnant, lactating, or of child bearing potential not using an adequate form of birth control
* Currently being treated with coumadin
* Forced vital capacity (FVC) <40% of predicted unless the tidal volume is > 600cc, as patients with significant bulbar weakness may show a falsely low FVC due to bulbar muscle spasticity

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Global impression of change by subject at eight weeks post injection

SECONDARY OUTCOMES:
Patient's subjective assessment of benefit
Change in volume of saliva produced over five minutes (measured with funnel and tube)
ALS Functional Rating Scale (ALSFRS)
Caregiver's subjective assessment of benefit
Change in anticholinergic medication doses and number of times per day suction is used
SEQOL-DW
Duration of benefit
Assessment of treatment assignment (final visit only)
Global assessment of change by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Carlayne E Jackson, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Charles B Simpson, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University of Kansas Medical Center/Neurology, 1008 Wescoe, Kansas City, Kansas
  - Carolinas MDA Neuromuscular/ALS Center; Carolinas Medical System; 1540 Garden Terrace, Charlotte, North Carolina